CLINICAL TRIAL: NCT06519357
Title: A Single-center, Self-controlled, Prospective Case Series Pilot Study to Assess the Effect of Lamivudine (3TC) on Neurocognitive Impairment Biomarkers and Type-I IFN (Interferon)-Stimulated Genes in the Plasma of Patients With Mild Cognitive Impairment (MCI)
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Fundación FLS de Lucha Contra el Sida, las Enfermedades Infecciosas y la Promoción de la Salud y la Ciencia (Other)
Collaborators: IrsiCaixa (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Lamiferon
Record Dates: First submitted 2024-07-19; First posted 2024-07-25 (Actual); Last update posted 2025-12-04 (Actual); Status verified 2025-06

CONDITIONS: Mild Cognitive Impairment
Keywords: Alzheimer; biomarkers
MeSH Terms: conditions — Cognitive Dysfunction | interventions — Lamivudine

STUDY DESIGN:
Intervention Model Description: Self-controlled, prospective case series pilot study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Lamivudine 300 (Other): Participants receive 300 mg of Lamivudine daily for 24 weeks
  Interventions: Drug: Lamivudine 300 MG

INTERVENTIONS:
Drug: Lamivudine 300 MG — Participants receive 300 mg of Lamivudine daily for 24 weeks

SUMMARY:
To assess the ability of lamivudine to lower the levels of neurocognitive impairment biomarkers in the plasma of patients with MCI and positive AD biomarkers in a 24 weeks-treatment period.

To assess the incidence, nature, and severity of Treatment Emergent Adverse Events (TEAE).

DETAILED DESCRIPTION:
To assess the ability of lamivudine to lower the levels of type-I IFN-stimulated genes in the plasma and cryopreserved PBMCs of patients with MCI and positive AD biomarkers in a 24 weeks-treatment period.

Exploratory objectives

To assess the ability of lamivudine to modify retrotransposons expression in cryopreserved PBMCs the plasma of patients with MCI and positive AD biomarkers in a 24 weeks-treatment period.

ELIGIBILITY:
Inclusion Criteria:

Male or female participants 55 to 90 years of age (both inclusive) at the time of signing the informed consent.

Diagnosis of prodromal AD: MCI due to AD according to National Institute on Aging-Alzheimer's Association (NIA-AA) criteria as determined by a neurologist, geriatrician, psychiatrist, or clinician approved by the Sponsor or designee.

Clinical Dementia Rating (CDR)-Global Score of 0.5

Imaging studies (MRI or CT) within 21 years prior to screening that exclude secondary causes of dementia.

that has findings consistent with AD and without any other disease that may cause dementia.

Documented confirmation of AD diagnosis by positive CSF AD signature or positive amyloid-PET AD signature. Amyloid positivityCSF AD positivity established with low levels of CSF Aβ1-42 or CSF Aβ1-42/Aβ1-40 and high levels of p-Tau. A CSF examination performed within 612 months prior to screening are is allowed. A positive amyloide-PET is defined as abnormal deposits of amyloid in the PET imaging. Subjects without documented positive AD biomarker status must have a positive CSF biomarker result from a sample provided at screening.

If receiving an approved medication for AD (i.e., donepezil, galantamine, rivastigmine, memantine, or memantine/donepezil combination product), must be on the medication with a stable dose for at least 4 weeks before the screening visit (dosing should remain stable throughout the study).

If receiving an OTC supplement for cognition (e.g., gingko biloba, omega-3 polyunsaturated fatty acid, vitamin E, curcumin), must not be exceeding the recommended dose and be at stable dose for at least 4 weeks prior to screening visit.

Able to visit the study center and undergo cognitive, functional, and other tests specified in the protocol.

Has a caregiver who:

Agrees to accompany the participant to all study visits and able to supervise the participant's compliance with the study procedures and provide detailed information about the participant.

Either lives with the participant or sees the participant on average for ≥ 1 hour/day ≥ 3 days/week, or in the Investigator's opinion, the extent of contact is sufficient to provide meaningful assessment of changes in participant behavior and function over time and provide information on safety and tolerability.

Can read, understand, and speak the designated language at the study center.

Caregiver must be cognitively able to fulfill the requirements of the study.

A male participant must agree to use a highly effective contraception method during the treatment period and for at least 3 months after the last dose of study treatment and refrain from donating sperm during this period.

A female participant is eligible to participate if she is not pregnant, not breastfeeding, and at least one of the following conditions applies:

Not a woman of childbearing potential (WOCBP) OR a WOCBP who agrees to use a highly effective contraception method during the treatment period and for at least 3 months after the last dose of study treatment.

A WOCBP must have a negative serum pregnancy test at screening and must use medically accepted means of contraception throughout the study.

Written informed consent provided by participant (or legal representative) and caregiver prior to any study-specific procedures.

Exclusion Criteria:

Any other cause of dementia shown by MRI or CT findings within 2 years of screening and neurological examination at screening.

Possible, probable, or definite vascular dementia according to the National Institute of Neurological Disorders and Stroke and Association Internationale pour la Recherché et l'Enseignement en Neurosciences (NINDS-AIREN) criteria.

Evidence of significant abnormality that would suggest another potential etiology for dementia (e.g., evidence of cerebral contusion, encephalomalacia, aneurysm, vascular malformation, > 10 microhemorrhages, macrohemorrhage, single infarct > 1 cm3).

Other central nervous system diseases that may cause cognitive impairment (e.g., cerebrovascular disease including cerebrovascular dementia, Parkinsonism, Huntington's disease, subdural hematoma, normal pressure hydrocephalus, brain tumor, Creutzfeldt-Jakob disease).

Concurrent or history of clinically significant psychiatric conditions (e.g., schizophrenia or bipolar affective disorder) that in the Investigator's opinion prevents the participant from participating or is likely to confound interpretation of drug effect or affect cognitive assessments.

Vitamin B12, folic acid, syphilis serology, and thyroid stimulating hormone (TSH) results that are thought to contribute to the severity of dementia or cause dementia. Participants may be enrolled if in the Investigator's medical judgment, the abnormal laboratory values are not the cause of the cognitive symptoms.

History of known or suspected seizures including febrile seizures (excluding self-limited childhood febrile seizures), a history of significant head trauma with loss of consciousness or recent unconsciousness that is not explained.

Acute or unstable cardiovascular disease, active peptic ulcer, uncontrolled hypertension, uncontrolled diabetes or any medical condition that may interfere with the completion of the clinical study.

Known allergies, hypersensitivity, or intolerance to lamivudine or similar products or excipients.

History of alcohol, substance abuse or dependence as per DSM-V criteria (except nicotine dependence) within the last 3 years.

Concurrent malignancies or invasive cancers diagnosed within the past 3 years except for non-metastatic basal cell carcinoma or squamous cell carcinoma of skin, in situ carcinoma of the uterine cervix or non-metastatic prostate cancer.

Sexually active WOCBP or man capable of fathering a child who do not consent to using medicinally acceptable contraception (such as surgical sterilization, intrauterine contraceptive device, condom, or diaphragm, an injectable or inserted contraceptive) during the study and for 3 months after the last dose of study treatment.

Use of anxiolytics, narcotics, or sleep aids in a manner that would interfere with cognitive testing, in the opinion of the investigator. Atypical antipsychotics may be used at the discretion of the Investigator. Tricyclic antidepressants and monoamine oxidase (MAO) inhibitors may be used at the discretion of the investigator.

Previous treatment with lamivudine.

Received an investigational product for AD within the last 3 months.

Participated in another clinical study within 4 weeks prior to this study.

Subject has any of the following laboratory findings at screening:

1. Severe liver dysfunction (Alanine aminotransferase > 2x upper limit of normal (ULN), aspartate aminotransferase > 2x ULN, or history of clinically significant liver disease in the investigator's judgment.
2. Hemoglobin ≤ 10 g/dl.
3. International Normalized Ratio (INR) > 1.5 or total bilirubin > 1.5 x ULN (unless subject has evidence of Gilbert's disease).
4. Renal impairment Creatinine clearance (CrCl) < 45 ml/min.
5. Poorly controlled diabetes as defined by hemoglobin A1C (HbA1C) > 8.
6. Positive blood screen for Human Immunodeficiency Virus (HIV-1 and 2), Hepatitis B surface antigen (HBsAg), or Hepatitis C virus antibodies (HCV-Ab) at Screening.

Body weight ≤ 35 kg.

Resides in a moderate to high dependency continuous care facility (residence in low grade assisted living facility where there is sufficient autonomy to permit valid evaluation of activities of daily living is allowed).

Any other reason that in the opinion of the investigator would make the participant ineligible to participate or to complete this study.

Refrain from donating blood or blood products from the screening visit until 3 months after the EOS/ET visit.

Ages: 55 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2024-10-28 (Actual); Primary Completion 2025-09-05 (Actual); Study Completion 2026-03 (Estimated)

PRIMARY OUTCOMES:
To assess the ability of lamivudine to lower the levels of neurocognitive impairment biomarkers in the plasma of patients with MCI and positive AD biomarkers in a 24 weeks-treatment period. | 24 weeks
  Percentage of change of pTau-217, total Tau, NfL, GFAP, Aβ42, Aβ40, and ratio in plasma from baseline visit to week 24 visit.
To assess the incidence, nature, and severity of Treatment Emergent Adverse Events (TEAE). | 48 weeks
  Safety and tolerability as measured by incidence, nature, and severity of treatment adverse events (AE), serious AE (SAE), and AE leading to withdrawal.

SECONDARY OUTCOMES:
To assess the ability of lamivudine to lower the levels of type-I IFN-stimulated genes in the plasma and cryopreserved PBMCs of patients with MCI and positive AD biomarkers in a 24 weeks-treatment period. | 24 weeks
  Fold change of type-I IFN-stimulated genes in plasma and cryopreserved PBMCs from baseline visit to week 24 visit.

CONTACTS AND LOCATIONS:
Locations (1):
- Germans Trias I Pujol Hospital, Badalona, BARCELONA, Spain

IPD SHARING:
Plan to Share IPD: No